CLINICAL TRIAL: NCT04244552
Title: A Phase 1b Dose Escalation and Expansion Trial to Investigate the Safety, Tolerability, Pharmacokinetics, and Biological Activity of ATRC-101 as Monotherapy and in Combination With Other Anticancer Agents in Adults With Advanced Solid Malignancies
Brief Title: A Phase 1b Trial of ATRC-101 in Adults With Advanced Solid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Atreca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATRC-101-A01
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Colorectal Cancer; Ovarian Cancer; Non-Small Cell Lung Cancer; Acral Lentiginous Melanoma; Head and Neck Squamous Cell Carcinoma; Hepatocellular Carcinoma; Esophageal Squamous Cell Carcinoma; Urothelial Carcinoma; DMMR Colorectal Cancer; MSI-H Colorectal Cancer; Melanoma; Platinum-Resistant Primary Peritoneal Carcinoma; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Epithelial Ovarian Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Hepatocellular; Esophageal Squamous Cell Carcinoma; Carcinoma, Transitional Cell; Melanoma; Triple Negative Breast Neoplasms | interventions — pembrolizumab; liposomal doxorubicin; 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ATRC-101 Q3W (Experimental)
  Interventions: Biological: ATRC-101
- ATRC-101 Q2W (Experimental)
  Interventions: Biological: ATRC-101
- ATRC-101 Q3W + Pembrolizumab (Experimental): Pembrolizumab 200mg IV Q3W or 400mg IV Q6W
  Interventions: Biological: ATRC-101; Biological: Pembrolizumab
- ATRC-101 Q2W + Pegylated liposomal doxorubicin (PLD) (Experimental): PLD 40mg/m^2 IV Run-in period of 28 days, and then 40mg/m^2 IV Q4W
  Interventions: Biological: ATRC-101; Drug: Pegylated liposomal doxorubicin (PLD)

INTERVENTIONS:
Biological: ATRC-101 — ATRC-101 is an engineered, fully-human IgG1 antibody derived from a naturally-occurring human antibody.
Biological: Pembrolizumab — Pembrolizumab (Keytruda®) is a humanized immunoglobulin G4 monoclonal antibody with high specificity of binding to the programmed cell death 1 (PD-1) receptor, thus inhibiting its interaction with programmed cell death ligand 1 (PD-L1) and programmed cell death ligand 2 (PD-L2).
  Arms: ATRC-101 Q3W + Pembrolizumab
Drug: Pegylated liposomal doxorubicin (PLD) — Pegylated liposomal doxorubicin (PLD) is doxorubicin hydrochloride (HCl), an anthracycline topoisomerase inhibitor that can bind DNA and inhibit nucleic acid synthesis. PLD is doxorubicin HCL encapsulated in liposomes formulated with surface-bound methoxypolyethylene glycol
  Other Names: DOXIL®, PLD
  Arms: ATRC-101 Q2W + Pegylated liposomal doxorubicin (PLD)

SUMMARY:
ATRC-101-A01 is a Phase 1b, open-label dose escalation and expansion trial of ATRC-101, an engineered fully human immunoglobulin G, subclass 1 (IgG1) antibody derived from a naturally occurring human antibody. The safety, tolerability, PK, and biological activity of ATRC-101 will be characterized when administered every two weeks (Q2W) or every 3 weeks (Q3W) as a monotherapy or in combination with other anticancer agents.

DETAILED DESCRIPTION:
For the monotherapy cohorts, including the efficacy expansion cohorts, enrollment is restricted to adults with inoperable, locally advanced or metastatic breast cancer, NSCLC, CRC, ovarian cancer, and acral melanoma, which are all tumor types that have demonstrated ATRC-101 immunoreactivity on at least 50% of tested commercially procured archival specimens.

For the pembrolizumab combination therapy cohort, enrollment is restricted to adults with inoperable, locally advanced or metastatic NSCLC, CRC (only MSI-H or dMMR), melanoma (with the exception of uveal melanoma), HCC, HNSCC, ESCC, UC or TNBC, that have been treated with anti-PD-1 or anti-PD-L1 therapy and have progressed radiographically or have achieved stable disease for a minimum of two months and who, in the judgment of their treating physicians, could benefit from a combination of ATRC 101 and pembrolizumab.

For the PLD combination therapy cohort, enrollment is restricted to adult females with inoperable, locally advanced or metastatic high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer that is platinum resistant, defined as progression during or within 6 months of the last dose of platinum-based chemotherapy OR breast cancer that is refractory to other standard therapies.

For target-enriched expansion cohorts, enrollment will be limited to participants with pretreatment tumor biopsies demonstrating ATRC-101 target expression above a predefined threshold by IHC at a central laboratory.

ELIGIBILITY:
Inclusion Criteria

* Confirmed diagnosis of:
* For the monotherapy cohorts: Inoperable, locally advanced or metastatic breast cancer, NSCLC, CRC, ovarian cancer, or acral melanoma that is refractory to standard therapy or for which no standard therapy exists. Participants who are considered intolerant of or ineligible for standard therapy(ies), as well as participants who have been offered but refused standard therapy(ies), may also be eligible.
* For the pembrolizumab combination therapy cohort: Inoperable, locally advanced or metastatic NSCLC, CRC (only MSI-H or dMMR), melanoma (with the exception of uveal melanoma), HCC, HNSCC, ESCC,UC, or TNBC with prior or ongoing anti-PD-1 or anti-PD-L1 treatment and have progressed radiographically or have achieved stable disease for a minimum of two months and who, in the judgment of their treating physicians, could benefit from a combination of ATRC-101 and pembrolizumab . The anti-PD-1/anti-PD-L1 therapy must be FDA approved for their cancer indication at the time of screening. Patients with the tumor types eligible for monotherapy that are TMB-H, MSI-H or dMMR and have had an unsatisfactory response to anti-PD-1/anti-PD-L1 therapy may enroll for the pembrolizumab combination, and additional indications that have been identified as ATRC-101 target positive and are FDA approved for pembrolizumab may be added following discussion with the study Medical Monitor.

  1. Individuals with BRAF mutant melanoma must have received BRAF inhibitors alone or in combination with a MEK inhibitor, if indicated.
  2. Individuals with NSCLC should have received platinum-based therapy unless contraindicated
* For the PLD combination therapy cohort: Inoperable, locally advanced or metastatic high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer that is platinum resistant, defined as progression during or within 6 months of the last dose of platinum-based chemotherapy OR breast cancer that is refractory to other standard therapies.
* Measurable disease based on RECIST 1.1, as assessed by the local site investigator/radiologist. As per RECIST, lesions situated in an area treated with radiation or other loco-regional therapy are considered measurable only if progression has been demonstrated in such lesions following loco-regional therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate organ and marrow function (i.e., without chronic, ongoing growth factor or transfusion support) at Screening as defined by the following laboratory parameters via central laboratory results:
* Absolute neutrophil count (ANC)

  1. For monotherapy and pembrolizumab combination therapy cohorts: ≥ 1000/µL
  2. For PLD combination therapy cohort: ≥ 1500/µL
* Platelet count ≥ 75,000/µL
* Hemoglobin ≥ 9.0 g/dL
* PT/INR, aPTT ≤ 1.5 x ULN unless participant is receiving a stable dose of therapeutic anticoagulation
* Albumin ≥ 3.0 g/dL
* Creatinine clearance or eGFR ≥ 30 mL/min as estimated by the Cockcroft-Gault equation
* AST/ALT ≤ 2 x ULN. If documented liver metastases, then ≤ 5X ULN
* Bilirubin

  1. For monotherapy and pembrolizumab combination therapy cohorts: ≤ 2 x ULN; or bilirubin ≤ 3 x ULN if due to Gilbert's or Crigler-Najjar disease
  2. For PLD combination therapy cohort: ≤ ULN
* Available representative tumor specimens in paraffin blocks (preferred) or ≥ 20 unstained slides (serial sections), with an associated pathology report, obtained after last systemic anticancer therapy and within 60 days prior to the planned first dose of investigational product (Cycle 1-Day 1). If fewer than 20 unstained slides are available, a discussion with the Medical Monitor is required prior to enrollment. If an archived sample is not available, participant must have a tumor that is amenable to biopsy without unacceptable risk of a major procedural complication and consent to have a tumor biopsy. Tumor lesions used for biopsy should not be lesions used as RECIST 1.1 target lesions unless there are no other lesions suitable for biopsy. If a RECIST target lesion is used for biopsy, the lesion must be ≥ 2 cm in longest diameter. Fine-needle aspirates, cell pellets from pleural effusions, ascites, and bone metastases are not acceptable.

  1. For the pembrolizumab combination therapy cohort: A biopsy collected within 60 days of the planned first dose of investigational product while the participant is receiving anti-PD-1/anti-PD-L1 therapy is acceptable.
  2. For target-enriched expansion cohorts, enrollment will be limited to participants with pretreatment tumor biopsies demonstrating ATRC-101 target expression above a predefined threshold by IHC at a central laboratory.
* Women of childbearing potential (WOCBP) and fertile males with partners who are WOCBP must use highly effective contraception (per CTFG 2014) from first dose and through 90 days after final dose of investigational product
* Willing and able to provide written informed consent and able to comply with all trial procedures

Exclusion Criteria

Individuals who meet any of the following criteria are not eligible to participate in this trial:

* Disease that is suitable for local therapy administered with curative intent.
* Malignant disease other than the malignancy to be investigated in this trial within the last 5 years with the exception of:

  a. malignancies previously treated with curative intent with a 5-year OS rate >90% (consultation with the Medical Monitor is required prior to enrollment).
* Autoimmune disease requiring systemic treatment (e.g., with disease modifying agents, corticosteroids, or immunosuppressive drugs) in the past 2 years. Hormone replacement therapy (e.g., insulin, thyroxine, and replacement-dose hydrocortisone) is not considered systemic treatment for the autoimmune disease.
* Active or prior paraneoplastic neurologic disorder of the central nervous system (CNS) or history of leptomeningeal disease
* Prior allogenic hematopoietic or solid organ transplant, including allogeneic cellular therapy (e.g., allogeneic chimeric antigen receptor (CAR)-modified T cells). Allogeneic bone grafts are not exclusionary.
* Clinically significant cardiovascular disease, e.g., cerebral vascular accident/stroke or myocardial infarction, within 6 months prior to first dose of investigational product, unstable angina, congestive heart failure (New York Heart Association ≥ Class III), or unstable cardiac arrhythmia requiring medication
* For the PLD Combination Therapy Cohort:

  1. Any history of documented congestive heart failure (CHF), arrhythmia, or uncontrolled hypertension (systolic BP > 200 mmHg or diastolic BP > 100 mmHg)
  2. Left ventricular ejection fraction measure by echocardiography or multigated radionuclide acquisition (MUGA) below normal limits for the institution
* Presence of active, symptomatic, or untreated CNS metastasis; or CNS metastasis that requires local directed therapy or increasing doses of corticosteroids within the 2 weeks prior to the planned first dose of investigational product. Individuals with treated and/or asymptomatic CNS disease may be enrolled if neurologically stable over the prior 2 weeks (and after consultation with the Medical Monitor) provided there is measurable disease (RECIST 1.1) outside of the CNS and there is no ongoing requirement for corticosteroids to manage the disease
* HIV infection with an AIDS-defining opportunistic infection within the past 12 months or with a CD4+ T cell count <350/µL
* Hepatitis B surface antigen (HbsAg) positive OR Hepatitis B core antibody (anti-HBc or HBcAb) positive and HBV viral load above the lower limit of quantification
* Hepatitis C antibody positive with HCV viral load greater than or equal to the lower limit of quantification
* Infection requiring intravenous antibacterial, antiviral, or antifungal therapy within 2 weeks prior to the planned first dose of investigational product
* Ongoing ≥ Grade 2 toxicity(ies) due to a previously administered anticancer agent with the following exceptions:

  1. Grade 2 neuropathy or alopecia
  2. For the monotherapy cohorts: Grade 2 immune-related endocrinopathy attributed to a checkpoint inhibitor and controlled with hormone replacement alone
* Treatment with biological agents (including monoclonal antibodies and cytokines) within 28 days of the planned first dose of investigational product with the following exception:

  a.For the pembrolizumab combination therapy cohort: -Anti-PD-1/anti-PD-L1 treatment within 28 days of the planned first dose of investigational product.
* Treatment with radiation, chemotherapy or anticancer small molecule therapy within 14 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. Treatment with nitrosoureas or mitomycin C require a 42-day washout prior to the planned first dose of investigational product
* For the PLD combination therapy cohort:

  1. Prior treatment with PLD
  2. Prior treatment with doxorubicin or other anthracycline at cumulative doses greater than 300mg/m2.

     1. Anthracycline equivalent doses: 1 mg Doxorubicin = 1.8 mg Epirubicin = 0.3 mg Mitoxantrone = 0.25 mg Idarubicin
  3. Anthracyclines or anti-HER2 agents, if last dose was administered < 1 year before enrollment
  4. Prior mediastinal irradiation > 3500 cGY
* Receipt of any investigational drug or device not otherwise specified above within 28 days or 5 half-lives (whichever is longer) prior to the planned first dose of investigational product
* Pregnant or breastfeeding; negative pregnancy status in WOCBP must be confirmed by serum pregnancy test at Screening
* History of ≥ Grade 3 infusion-related reaction associated with antibody administration, or:

  1. For the monotherapy cohorts: Known allergy/intolerance to ATRC-101 or its excipients
  2. For the pembrolizumab combination therapy cohort: Known allergy/intolerance to ATRC-101, anti-PD-1 or anti-PD-L1, , or their excipients
  3. For the PLD combination therapy cohort: Known allergy/intolerance to ATRC-101, doxorubicin, or to the excipients of ATRC-101 or PLD
* Major surgery or significant traumatic injury occurring within 28 days prior to the planned first dose of investigational product. If major surgery occurred > 28 days prior to Cycle 1-Day 1, individual must have recovered adequately from the toxicity and/or complications from the intervention prior to Cycle 1-Day 1
* Prior treatment with ATRC-101
* Intercurrent illness that is either life-threatening or of clinical significance such that it might limit compliance with trial requirements, or in the Investigator's assessment would place the participant at an unacceptable risk for participation. Uncontrolled pleural effusion, pericardial effusion or ascites requiring recurrent drainage procedures is exclusionary
* Receipt of a live, attenuated vaccine within 28 days of planned Cycle 1-Day 1. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed. Intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed. Replication-incompetent viral, mRNA, subunit, conjugate, and toxoid vaccines are allowed.
* COVID-19 (SARS-CoV-2) pandemic consideration: The COVID-19 vaccination should not be delayed; however, caution should be exercised when combining vaccination with cancer therapy, particularly immunotherapy. The COVID-19 vaccines can cause transient lymphadenopathy and potentially impact assessment of disease burden during screening and/or on-study. To allow correct interpretation and reduce equivocal findings, investigators should discuss with the participant appropriate timing and selection of anatomic site of vaccination (alternative) with respect to imaging scans (MRI or CT). Screening scans should be acquired before the first dose of a COVID-19 vaccine or 4-6 weeks after the second dose of the vaccine. Because cancer patients are considered vulnerable population, after COVID-19 vaccination there is also a potential for heightened immune related adverse events including CRS. Investigators should use judgement when evaluating and managing potentially overlapping adverse events and in establishing causality with the study treatment (Schönrich and Raftery 2019; Desai et al. 2021; Edmonds et al. 2021; Indini et al. 2021)

For the pembrolizumab combination therapy cohort ONLY:

* Experienced ≥ Grade 3 immune related adverse events while on immunotherapy prior to enrollment
* Have not recovered from Grade 2 immune related adverse events attributed to immunotherapy to Grade 1 or baseline prior to enrollment.
* NSCLC with epidermal growth factor receptor (EGFR) or anaplastic lymphoma receptor tyrosine kinase (ALK) genomic tumor alterations
* Isolated intracranial relapse
* Interstitial lung disease or active, non-infectious pneumonitis
* Signs and symptoms consistent with clinically significant, decreased pulmonary function: (1) blood saturation oxygen level (SpO2) < 90% at rest on room air; (2) dyspnea at rest (CTCAE v. 5.0 ≥ Grade 3) or supplemental oxygen used to maintain adequate oxygenation within 14 days prior to the planned first dose of investigational product
* Ongoing immune-related toxicity or immune-related toxicity requiring systemic corticosteroids for 30 or more consecutive days for a prior immune related adverse event before initiation of study treatment

For the PLD combination therapy cohort ONLY:

•Prior drug-induced cardiotoxicity, defined as a sustained decrease in the ejection fraction (EF) of > 15%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of DLTs (dose escalation cohorts only), treatment emergent adverse events (TEAEs), and changes in safety parameters | 24 months

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of ATRC-101 | 24 months
Elimination half-life (t1/2) of ATRC-101 | 24 months
Area under the plasma concentration-time curve from zero to the last measurable concentration [AUC(0-t)] of ATRC-101 | 24 months
Incidence of anti-drug antibodies (ADAs) and ATRC-101 neutralizing antibodies | 24 months
Overall Response Rate (ORR), defined as the proportion of participants with a CR or a PR on two consecutive occasions > 4 weeks apart, according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | 24 months
Enumeration of tumor-infiltrating CD8+ lymphocytes (TILs) in tumor biopsy specimens at baseline and during treatment | 24 months
Distribution of tumor-infiltrating CD8+ lymphocytes (TILs) in tumor biopsy specimens at baseline and during treatment | 24 months
Levels of ATRC-101 immunoreactivity expressed as H-score, tumor proportion score, and maximum intensity | 24 months
For the PLD Combination Therapy Cohort: ATRC-101 immunoreactivity in tumor biopsies at baseline and during treatment | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Khurana, PhD, Study Director — Atreca, Inc.
Locations (19):
- United States (19):
  - Mayo Clinic, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles Hematology/Oncology, Los Angeles, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Florida Cancer Specialists, Lake Mary, Florida
  - University of Miami Hospital - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Carolina BioOncology, Huntersville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Stephenson Cancer Center, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Oncology Consultants, PLLC, Houston, Texas

IPD SHARING:
Plan to Share IPD: No